CLINICAL TRIAL: NCT03832946
Title: A Randomized, 52 Week, Double-blind, Multicentre, Parallel, Placebo-controlled Phase 2b Study in Subjects With Idiopathic Pulmonary Fibrosis (IPF) Investigating the Efficacy and Safety of GB0139, an Inhaled Galectin-3 Inhibitor.
Brief Title: A Study to Test the Efficacy and Safety of Inhaled GB0139 in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galecto Biotech AB (Industry)
Collaborators: Syneos Health (Other); bioRASI, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GALACTIC-1; 2018-002664-73 (EudraCT Number)
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-04

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
Keywords: TD139; Idiopathic pulmonary fibrosis; Galectin-3 inhibitor; GB0139
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — GB-0139

STUDY DESIGN:
Intervention Model Description: All subjects eligible for the study will be randomised into one of the two treatment arms:
  A. GB0139 3 mg once a day B. Placebo once a day
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is a double-blind study. The blinding will be maintained throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A. GB0139 3 mg once a day (Experimental): Inhalation of GB0139
  Interventions: Drug: GB0139
- B. Placebo once a day (Placebo Comparator): Inhalation of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GB0139 — GB0139 is a galectin-3 inhibitor designed to modulate the fibrogenic response to tissue injury. It is administered as inhalation once a day.
  Other Names: TD139
  Arms: A. GB0139 3 mg once a day
Drug: Placebo — Placebo is administered as inhalation once a day
  Arms: B. Placebo once a day

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase 2b trial in subjects with IPF (idiopathic pulmonary fibrosis) investigating the efficacy and safety of GB0139.

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy and safety of GB0139, a galectin-3 inhibitor, administered by dry powder inhalation over 52 weeks. GB0139, given once per day, will be compared to placebo. GB0139 was previously known as TD139.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged ≥ 40 years of age with a diagnosis of IPF established during the previous five years according to ATS/ERS/Fleischner criteria.
2. Lung function parameters as follows:

   1. Forced Vital Capacity (FVC) > 45% of the predicted value at screening
   2. Diffusion lung capacity for carbon monoxide (DLCO) (corrected for Hb) of 30% to 79% of the predicted value at screening
3. Subjects who currently are not being treated with nintedanib or pirfenidone; or cannot tolerate nintedanib or pirfenidone
4. Subjects must sign and date a written, IRB/EC approved informed consent form and any required authorization prior to initiation of any study procedures.

Exclusion Criteria:

1. Currently has significant airways obstruction: Forced Expiratory Volume in 1 s (FEV1)/Forced Vital Capacity (FVC) ratio of < 0.7 at screening.
2. Has clinical evidence of active infection, including, but not limited to, bronchitis, pneumonia, sinusitis, urinary tract infection, and cellulitis.
3. Has a history of malignancy within the last 2 years with the exception of basal cell carcinoma, chronic lymphocytic leukaemia (under observation) and prostate cancer requiring anti-androgens, localised treatment (minor surgery, radiotherapy) and/or managed by observation.
4. Has any condition other than IPF that, in the opinion of the investigator, is likely to result in the death of the subject within the next 2 years.
5. Presence of other disease that may interfere with testing procedures or in the judgement of the Investigator may interfere with trial participation or may put the patient at risk when participating in this trial.
6. Is likely to receive lung transplantation within the next 12 months.
7. Currently receiving nintedanib, pirfenidone, high dose corticosteroid, cytotoxic (e.g., chlorambucil, azathioprine, cyclophosphamide, methotrexate), vasodilator therapy for pulmonary hypertension (e.g., bosentan). A current dose of less than or equal to 15 mg/day of prednisone or its equivalent is acceptable if the dose is anticipated to remain stable during the study.
8. Prior use of GB0139 (also called TD139) or previously randomized in GALACTIC-1.
9. Prior use of nintedanib or pirfenidone within 7 days of initiation of screening.
10. Prior use of investigational drugs within 30 days (or 5 half-lives, whichever is longer) of initiation of screening.
11. Participating in another clinical trial, either interventional or observational.
12. Has a history of unstable or deteriorating cardiac or pulmonary disease (other than IPF) within the previous six months, including, but not limited to, the following:

    1. Unstable angina pectoris or myocardial infarction, or percutaneous coronary intervention within the last 6 months
    2. Congestive heart failure requiring hospitalization
    3. Uncontrolled clinically significant arrhythmias
13. If female, the subject is pregnant or lactating or intending to become pregnant before participating in this study during the study and within (5 half- lives plus 30 days) after last dose of the study drug; or intending to donate ova during such time period.
14. Woman considered to be of childbearing potential who do not use highly effective birth control methods during the study.
15. Hypersensitivity to the active substance (TD139/GB0139) or the excipient (lactose).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toby Maher, MD, PhD, Principal Investigator — Keck Medicine of USC
Locations (128):
- United States (34):
  - SEC Clinical Research, Andalusia, Alabama
  - Jasper Summit Research, LLC Pulmonary & Sleep Associates, Jasper, Alabama
  - Palmtree Clinical Research Inc, Palm Springs, California
  - Paradigm Research, Redding, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Health Shands Hospital, Gainesville, Florida
  - Harmony Medical Research Institute, Inc, Hialeah, Florida
  - Advanced Research for Health Improvement, Naples, Florida
  - Broward Research Centre, Pembroke Pines, Florida
  - Avanza Medical Research Centre, Pensacola, Florida
  - Coastal Pulmonary Critical Care PLC, St. Petersburg, Florida
  - Tampa General Hospital/Uni Florida, Tampa, Florida
  - Piedmont Healthcare Pulmonary and Critical Care Research, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - DC Research Works, Marietta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - LaPorte County Institute for Clinical Research, Michigan City, Indiana
  - University of Kansas Medical Centre, Kansas City, Kansas
  - University of Louisville Hospital, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Harvard Medical School - Brigham and Womens Hospital (BWH), Boston, Massachusetts
  - The Lung Research Center LLC, Chesterfield, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Pulmonlx LLC, Greensboro, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Centre at Houston, Houston, Texas
  - University of Texas Health Sciences Center at Houston, Houston, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - University of Utah Health Scieces Center, Salt Lake City, Utah
  - TPMG Clinical Research, Williamsburg, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - Lung Research QLD, Chermside, Queensland
  - Flinders Medical Centre, Adelaide, South Australia
  - Respiratory Clinical Trials, Kent Town, South Australia
  - Institute for Respiratory Health Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - TrialsWest, Spearwood, Western Australia
- Belgium (5):
  - Cliniques Universitaires St-Luc, Louvain-la-Neuve, Wallon Region
  - UZ Antwerp, Antwerp
  - CUB Hopital Erasme, Brussels
  - UZ Leuven- Campus Gasthuisberg, Brussels
  - CHU UCL Namur site Godinne, Namur
- Canada (4):
  - Firestone Institute for Respiratory Health, Hamilton, Ontario
  - Dr Anees Medicine Professional Corporation, Windsor, Ontario
  - Dr Dhar Medical Practice, Windsor, Ontario
  - Toronto General Hosp Research Inst, Toronto
- France (10):
  - Groupe Hospitalier Hopitaux Universitaires Paris-Seine-Saint-Denis-Hopital Avicenne, Bobigny
  - CHRU Lille - Hopital Calmette, Lille
  - Hopital Nord de Marseille, Marseille
  - APHP - Hopital Europen Georges-Pompidou, Paris
  - Hopital Bichat, Paris
  - Centre Hospitalier Universitaire de Rennes Hopital Pontchaillou, Rennes
  - CHU de la Réunion Site SUD (Terre Sainte), Saint-Pierre
  - CHU de la Réunion- Site Félix Guyon, Saint-Pierre
  - Hopitaux Universitaires de Strasborg Service de Pneumologie Nouvel Hopital Civil, Strasbourg
  - Centre Hospitalier Rgional et Universitaire - Hopital Bretonneau, Tours
- Georgia (2):
  - Chapidze Emergency Cardiology Center, Tbilisi
  - The First Medical Center, Tbilisi
- Germany (11):
  - Thoraxklinik-Heidelberg gGmbH, Heidelberg, Baden-Wurttemberg
  - Lungenfachklinik Immenhausen Department for Clinical Studies, Immenhausen, Hesse
  - ZMS Zentrum für medizinische Studien GmbH, Warendorf, Rhine-Westphalia
  - Klifeck GmbH Praxis Med. Gerald Eckhardt, Delitzsch, Saxony
  - Studienzentrum Dr.med Falk Brunner FA fuer Innere Medizin und Pneumologie, Leipzig, Saxony
  - CIMS Studienzentrum Bamberg GmbH, Bamberg
  - Krankenhaus Donaustauf, Donaustauf
  - Ruhrlandklinik Essen, Essen
  - Universitaetsklinikum Leipzig Klinik und Poliklinik für Onkologie, Gastroenterologie, Hepatologie, P, Leipzig
  - POIS Leipzig GbR, Leipzig
  - Klinikum Grossadern der Ludwig-Maximilians-Universitaet Muenchen, Munich
- Trinity Centre for Health Sciences, Dublin, Ireland
- Israel (5):
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kefar Sava
  - Pulmonary Institute Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
- Italy (9):
  - University-Hospital Policlinico Vittorio Emanuele, Catania
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Giuseppe Clinica Malattie dell Apparato Respiratorio, Milan
  - University Hospital of Mondena-AOU - Policlinico di Modena, Modena
  - A.O. Dei Colli OSPEDALE MONALDI, Napoli
  - Ospedale GB Morgagni, Padua
  - Istituto Mediterraneo Trapianti e Terapia Alta Specializzazione (ISMETT), Palermo
  - Azienda Ospedaliera Universitaria Senese, Siena
  - AOU Città della Salute e della Scienza, PO Molinette, Turin
- Poland (5):
  - Oddział Kliniczny Pulmonologii i Alergologii Szpitala Uniwersyteckiego w Krakowie, Krakow, Lesser Poland Voivodeship
  - Instytut Gruzlicy i Chorob Pluc, I Klinika Chorob Pluc, Warsaw, Masovian Voivodeship
  - Klinika Alergologii Pneumonologii, Gdansk, Pomeranian Voivodeship
  - Szpital Kliniczny Przemienienia Pańskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Uniwersytecki Szpital Kliniczny Nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz, Łódź Voivodeship
- Russia (8):
  - Regional Clinical Hospital No. 3, Chelyabinsk
  - Kazan SMU, Republican Clinical Hospital of MOH, Republic of Tatarstan, Kazan'
  - OLLA-MED, Moscow
  - Pulmonology Scientific Research Institute, Moscow
  - Evdokimov Moscow State University of Medicine and Dentistry, Moscow
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - Soloviev Clinical Emergency Hospital, Yaroslavl
  - LLC "Medical Association Novaya Bolnitsa", Yekaterinburg
- Spain (11):
  - Hospital Univ. Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Lucas Augusti, Lugo, Galicia
  - Hospital Universitario Quiron Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Policlinica Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hopital de Bellvitge, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital General de Valencia, Valencia
- Ukraine (5):
  - Chernivtsi Regional Clinical Hospital, Chernivtsi
  - National Institute of Phthisiology and Pulmonology n.a. F.G.Yanovsky, Kyiv
  - National Research Centre for Radiation Medicine of The National Academy of Medical Sciences of UKR, Kyiv
  - Ternopil Municipal City Hosipital 2, Ternopil
  - Medical Centre Pulse, Vinnytsia
- United Kingdom (13):
  - Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire
  - Royal Devon and Exeter Hospital, Exeter, Devon
  - Royal Brompton Hospital, London, Greater London
  - Wythenshawe Hospital, Manchester, Greater Manchester
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Glenfield Hospital, Leicester, Leicestershire
  - Aintree Unversity Hospital NHS Foundation Trust, Liverpool, Merseyside
  - Newcastle Royal Victoria Infirmary, Newcastle upon Tyne, Newcastle
  - Nottingham City Hospital, Nottingham, Nottinghamshire
  - Sheffield Teaching Hospitals NHS Foundation Trust - Royal Hallamshire Hospital (RHH), Sheffield, South Yorkshire
  - Birmingham Heartlands Hospital, Birmingham, West Midlands
  - Clinical Research Centre - Respiratory North Bristol NHS Trust Southmead Hospital, Bristol
  - Royal Infirmary of Edinburgh, Edinburgh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rebelo AL, Chevalier MT, Russo L, Pandit A. Role and therapeutic implications of protein glycosylation in neuroinflammation. Trends Mol Med. 2022 Apr;28(4):270-289. doi: 10.1016/j.molmed.2022.01.004. Epub 2022 Feb 1. PMID 35120836
- [Derived] Park AM, Khadka S, Sato F, Omura S, Fujita M, Hsu DK, Liu FT, Tsunoda I. Galectin-3 as a Therapeutic Target for NSAID-Induced Intestinal Ulcers. Front Immunol. 2020 Sep 23;11:550366. doi: 10.3389/fimmu.2020.550366. eCollection 2020. PMID 33072090

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A. GB0139 3 mg Once a Day | B. Placebo Once a Day
Started | 102 | 70
Completed | 55 | 38
Not Completed | 47 | 32
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Change in Protocol forbidding use of Nintedanib / Pirfenidone | 30 | 22
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 12 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A. GB0139 3 mg Once a Day | B. Placebo Once a Day | Total
Number analyzed (Participants) | 102 | 70 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (7.59) | 71.7 (7.36) | 72.176 (7.48)
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical: <70 | 34 | 26 | 60
  Age, Categorical: >=70 | 68 | 44 | 112
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 22 | 49
  Male | 75 | 48 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 5
  Not Hispanic or Latino | 95 | 63 | 158
  Unknown or Not Reported | 7 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 98 | 69 | 167
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48
  Ukraine | 4 | 2 | 6
  United Kingdom | 27 | 15 | 42
  Spain | 1 | 4 | 5
  Canada | 1 | 1 | 2
  Ireland | 1 | 1 | 2
  Poland | 6 | 5 | 11
  Italy | 1 | 2 | 3
  Georgia | 8 | 1 | 9
  Israel | 10 | 5 | 15
  Australia | 8 | 1 | 9
  France | 4 | 3 | 7
  Germany | 2 | 4 | 6
  Russia | 6 | 2 | 8
Forced Vital Capacity (FVC) in mL [Mean (Standard Deviation); unit: mL] | 3003.1 (861.58) | 2859.1 (876.13) | 2944.5 (867.88)

OUTCOME MEASURES:

1. Primary Outcome: Annual Rate of Decline in Forced Vital Capacity (FVC)
Description: Efficacy of GB0139 as measured by the annual rate of decline in FVC expressed in mL
Time Frame: 52 weeks
Measure: Mean (95% Confidence Interval); unit: mL/Year
Arm/Group | A. GB0139 3 mg Once a Day | B. Placebo Once a Day
Number analyzed (Participants) | 100 | 68
mL/Year | -316.60 [-394.86 to -238.35] | -127.41 [-221.12 to -33.71]

2. Secondary Outcome: Number of Participants With Respiratory Related Hospitalizations
Description: Number of Participants with Respiratory Related Hospitalizations from randomisation (including acute exacerbation of IPF).
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | A. GB0139 3 mg Once a Day | B. Placebo Once a Day
Number analyzed (Participants) | 102 | 70
Participants | 17 | 5

3. Secondary Outcome: Assessment of Respiratory Related Quality of Life Using the St. George's Respiratory Questionnaire (SGRQ)
Description: Change from baseline to WK52 in the SGRQ total score. The SGRQ is a 50-item questionnaire split into three domains: symptoms, activity and impact. Weighting of both individual domains and the total score produces a range from 0 to 100, with higher scores indicating a poorer health-related quality of life.
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A. GB0139 3 mg Once a Day | B. Placebo Once a Day
Number analyzed (Participants) | 68 | 48
score on a scale | 4.201 (20.0648) | -4.77 (14.7286)

ADVERSE EVENTS:
Time Frame: 52 weeks (Includes all AEs with a start date up to and including Day 379 (52 weeks + 14 days)
Arm/Group | A. GB0139 3 mg Once a Day | B. Placebo Once a Day
All-Cause Mortality (participants affected / at risk) | 8/102 | 5/70
Serious Adverse Events (participants affected / at risk) | 24/102 | 11/70
Other Adverse Events (participants affected / at risk) | 80/102 | 50/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A. GB0139 3 mg Once a Day (N=102) | B. Placebo Once a Day (N=70)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 4 (4) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Septic Shock (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0)
Localised Infection (Infections and infestations) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1)
Necrosis (General disorders) | 1 (1) | 0 (0)
Sudden Death (General disorders) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine tumour of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Abdominal Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cerebral microangiopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Pernicious anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A. GB0139 3 mg Once a Day (N=102) | B. Placebo Once a Day (N=70)
Lower Respiratory Tract Infection (Infections and infestations) | 12 (19) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 4 (4)
Nasopharyngitis (Infections and infestations) | 4 (7) | 3 (4)
Bronchitis (Infections and infestations) | 6 (8) | 3 (4)
Urinary Tract Infection (Infections and infestations) | 5 (8) | 1 (2)
Tooth Abcess (Infections and infestations) | 3 (3) | 0 (0)
Tooth Infection (Infections and infestations) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1) | 1 (1)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Coronavirus Infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Oral Herpes (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Root Canal Infection (Infections and infestations) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (24) | 9 (9)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sputum Increased (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sputum Discoloured (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 4 (4) | 2 (2)
Asthenia (General disorders) | 4 (4) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Malaise (General disorders) | 1 (2) | 0 (0)
Vaccination Site Pain (General disorders) | 1 (2) | 0 (0)
Feeling Cold (General disorders) | 1 (1) | 0 (0)
Influenza Like Illness (General disorders) | 1 (1) | 0 (0)
Vaccination Site Rash (General disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb Mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (13) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (6) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 7 (7) | 2 (5)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Essential Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Mental Impairment (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Sensory loss (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial hypoxia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Gout (Metabolism and nutrition disorders) | 2 (3) | 1 (2)
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Folate Deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Increased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (5) | 0 (0)
Vaccination Complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (3)
Limb Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eyelid contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Soft Tissue Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weight Decreased (Investigations) | 4 (4) | 3 (3)
Forced vital capacity decreased (Investigations) | 2 (2) | 2 (2)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Monoclonal Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Epiretinal membrane (Eye disorders) | 0 (0) | 1 (1)
Episcleritis (Eye disorders) | 0 (0) | 1 (1)
Eye haematoma (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 2 (2)
Autoimmune disorder (Immune system disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatic atrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 5 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
COVID-19 (Infections and infestations) | 13 (14) | 3 (4)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Localised Infection (Infections and infestations) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 5 (5)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigators must agree to maintain the confidentiality of the study at all times and must not reveal any information relating to the study without express permission from the study Sponsor.

DOCUMENTS (2):
  • Study Protocol (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT03832946/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT03832946/SAP_001.pdf